CLINICAL TRIAL: NCT00781781
Title: Multicenter, Openlabel, Phase II Intergroups (GELTAMO/GETH) Trial, on the Use of Alemtuzumab for Unrelated Donor Reduced Intensity Conditioning Allogenic Transplant in Hematological Malignancies Patients
Brief Title: Alemtuzumab Use (MabCampath®) in Hematopoietic Transplant of Unrelated Donor With Reduced Intensity Conditioning
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit the number of patients established in the study protocol (34 of 40)
Sponsor: CABYC (Industry)
Collaborators: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALOTIRNE-EC06007; 2007-006440-22 (EudraCT Number)
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2008-10

CONDITIONS: Graft Versus Host Disease
Keywords: Myeloid and Lymphoid malignances
MeSH Terms: conditions — Graft vs Host Disease | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): High risk patients (at least one GVHD high risk criterion):
  Total dose 100 mg in 5 doses of 20 mg, days -8 to -4 (inclusive).
  Interventions: Drug: Alemtuzumab
- 2 (Experimental): Low Risk patients (no GVHD high risk criterion):
  Total dose 50 mg inn 5 dosing OF 10 mg, days -5 to -1 (inclusive).
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — High risk: Total dose 100 mg in 5 doses of 20 mg, days -8 to -4 (inclusive) Low risk: Total dose 50 mg inn 5 dosing OF 10 mg, days -5 to -1 (inclusive).
  Other Names: MabCampath

SUMMARY:
The purpose of this study is to analyze the results of incidence and severity of acute and chronic GVHD, (see addendum II) and of disease free survival with Alemtuzumab use (MabCampath®) in haematopoietic transplant of unrelated donor with reduced intensity conditioning.

DETAILED DESCRIPTION:
Each patient will be assigned to one of the two dosing schedules and total dose of drug envisaged in the study. The assignation to conventional or reduced Alemtuzumab (MabCampath) dose will be done depending on the age and risk of suffering GVHD, in function of variables coming from general experience.

High risk of GVHD criteria:

Gender incompatibility: male patient of female donor. HLA incompatibility: non identical high resolution typing in HLA A, B, C, DRB1, DQB1 (identity less than 10/10 alleles by high resolution) Age of patient more or equal than 55 years

Conventional doses in high risk (at least one criterion of GVHD high risk):

100 mg de Alemtuzumab IV total dose in 5, 20 mg fractions, days -8, -7, -6, -5 and -4.

Reduced dose in low risk cases (no criteria of GVHD high risk):

50 mg de Alemtuzumab IV total dose en 5 fractions of 10 mg, days -5, -4, -3, -2 and -1.

ELIGIBILITY:
Inclusion criteria:

* Patients with haematological or lymphoid malignancies with allogenic transplantation indication:

  * High risk follicular NHL, mantle HHC and other low grade NHC (e.g lymphoplasmacytic, extranodal or from marginal zone).

    1. Disease that does not obtain a CR with Fludarabine or antiCD-20 including chemotherapy.
    2. Relapse after autologous transplant.
    3. Non candidates to autologous transplant in 2nd CR (e.g. mobilization failure, or persistent marrow infiltrate).
  * Poor prognosis chronic lymphoblastic leukaemia (CLL): Del 11q, Del 17p, complex cariotype; B symptoms, progressive low cell count by marrow infiltration, lymphocytosis or enlarged lymph nodes, or progressive spleen growth.
  * High grade lymphoma transformed from a low grade non Hodgkin's lymphoma or from a chronic lymphocitic leukaemia
  * High risk T peripheral lymphoma, with IPI > or = 2, non susceptible of autologous transplant, or relapsed after autologous transplant
  * Primarily refractory high risk Hodgkin's disease, relapse in patients not susceptible of autologous transplant or relapse after autologous transplant.
  * High risk acute mieloblastic leukaemia (AML) in 1st CR, or AMC > or = 2 CR, including AML after MDS and secondary AML.
  * High risk acute lymphoblastic leukaemia (ALL) because of poor response to induction chemotherapy (>10% blasts day +14 or no RC day +28-35), or by cytogenetic criteria: Ph+ or 11q23.
  * High risk myelodisplastic syndromes (SMD) type RAEB-1 or AREB-2 with IPSS >Int-1.
* For the inclusion in transplant patients with ALL or AML must be in CR, patients with MDS must have <10% blasts en la BM, and patients with lymphoid malignancies must show previous chemosensitivity, with PR or CR.
* Patients 40 to 65 years old. Patients outside this age range could be included according to participating centres criteria.
* Patients in the study population lacking a compatible related donor, and with a possible compatible unrelated donor (>=9/10 by 10 alleles high resolution typing: HLA-A, B, C, DRB1, DQB1) to assign the patients to a risk in subgroup.
* Signed informed consent.
* Not fulfilling any of the following exclusion criteria.

Exclusion Criteria:

* Liver (≥ x3 UNL), kidney (GF <40ml/min), cardiac (LVEF <40%) or respiratory (DLCO & FVC <40% of expected) function tests impairment.
* HIV injection.
* Absence of signed informed consent.
* Progressive disease previous to transplant or not fulfilling the above mentioned response criteria.
* Other co-morbidities that contraindicate CT.
* Pregnant and/or breast-feeding women or with pregnancy risk by inadequate contraception.
* Life expectancy <6 months.
* Mental or psychiatric deficiency impeding adequate understanding and consent to therapy
* Hypersensitivity as shown by anaphylactic reaction to any of the DRUGS used in the trial.
* Active infectious process.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Analyze the results of incidence and severity of acute and chronic GVHD | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Duarte, MD, Ph.D, Study Director — ICO Bellvitge. Hospital Duran i Reynals
Locations (10):
- Spain (10):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - Vall de Hebron, Barcelona, Barcelona
  - ICO Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic i Provincial., Barcelona, Catalonia
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Morales Meseguer, Murcia, Murcia
  - Hospital Clinico de Valencia, Valencia, Valencia